CLINICAL TRIAL: NCT03866915
Title: Validity of Aortic Pulse Wave Velocity in Predicting the 6- Minute Walking Test Before Major Non-cardiac Surgery (6WAVE)
Brief Title: Validity of Aortic Pulse Wave Velocity in Predicting the 6- Minute Walking Test Before Major Non-cardiac Surgery
Acronym: 6WAVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Responsible Party: Sponsor
Other Study IDs: REDGERM06
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Perioperative/Postoperative Complications; Surgery; Exercise Tolerance
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective surgery: All patients older than 18 years undergoing elective surgery that receive a preoperative visit by anesthesiologists in which Aortic pulse wave velocity measurement and the 6 minutes walking test (6MWT) is carried out
  Interventions: Diagnostic Test: Aortic pulse wave velocity measurement; Diagnostic Test: 6 minutes walking test

INTERVENTIONS:
Diagnostic Test: Aortic pulse wave velocity measurement — Aortic pulse pulse wave velocity (AoPWV) measured by photoplethysmography
Diagnostic Test: 6 minutes walking test — This test is performed routinely in the pre-rehabilitation units or in external anesthesiology consultations during the preoperative visit. In essence, it consists in measuring the maximum distance the patient is able to walk in 6 minutes, in a short walk in a corridor, simultaneously assessing the heart rate, oxygen saturation and the degree of dyspnea. In general, healthy people can walk between 400 and 700 meters in 6 minutes, depending on age, height and sex.
  Other Names: 6MWT

SUMMARY:
Methods: Prospective observational study in adult patients requiring preoperative evaluation

Objectives: To determine the correlation between the aortic pulse wave velocity (AoPWV) and the distance walked in the 6-minute walk test (6MWT) Sample Size: For a desired precision of estimate of ± 0.10 (95% confidence interval) around a postulated validity correlation coefficient of r = 0.70 (for an AoPWV in the distance prediction of 6MWT) a sample of 100 patients. By allowing a 25% wear rate, a final sample size of 125 participants is required Inclusion criteria: Patients older than 18 years undergoing any surgery and who require pre-anesthesia Statistical analysis If the variables have a normal distribution, the Pearson correlation coefficient (r2) is used, which is between -1 and 1. Where -1 indicates the highest possible negative linear relationship (increasing the value of a variable decreases the another), 0 that there is no association, +1 positive correlation. From 0.7 negative or positive, it is said that the association is strong.

Linear regression models of ordinary least squares will be applied to obtain the validity coefficient (r) and the standard error of the estimate (SEE): the typical error associated with the prediction the AoPWV with the distance traveled in the 6MWD test in each individual patient. The analysis of the receiver operating characteristic curve (ROC) will be used to derive cutoff points for an AoPWV value for the prediction of a 6MWD less than 427 meters

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years undergoing elective surgery that receive a preoperative visit by anesthesiologists.

Exclusion Criteria:

* Patients undergoing emergency surgery

  * Patients under 18 years of age
  * Patients who refuse to participate
  * Patients unable to perform the 6MWT
  * Claudication of the lower extremities and inability to maintain a constant pace of walking on level ground

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
AoPWV validity: relationship between AoPWV and 6MWT distance | 1 day
  The validity of AoPWV-physiological parameter measured non-invasively by photoplethysmography-will be evaluated to predict the distance traveled in 6MWT in adult patients undergoing any type of elective surgery

SECONDARY OUTCOMES:
AoPWV threshold | 1 day
  AoPWV threshold associated with a 6MWD threshold of 427 meters that defines the patient at risk

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ripollés Melchor, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; Ane Abad Motos, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; José M Ramírez, Study Chair — Lozano Blesa University Hospital, Zaragoza, Spain; César Aldecoa, Study Chair — Río Hortega University Hospital, Valladolid, Spain
Locations (3):
- Spain (3):
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided